CLINICAL TRIAL: NCT00122486
Title: Phase 2 Study of Tenofovir Disoproxil Fumarate (TDF) for Prevention of HIV
Brief Title: Study of Tenofovir Disoproxil Fumarate (TDF) for Prevention of HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FHI 360 (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9780
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2006-08-01 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate

SUMMARY:
This Phase 2 study involving tenofovir disoproxil fumarate (TDF) will assess the extended safety of TDF 300 mg per day among young women who are not HIV-infected.

DETAILED DESCRIPTION:
The protocol describes a randomized, fully-masked, parallel, placebo-controlled study of TDF for pre-exposure prophylaxis of HIV in high-risk women. TDF was selected for investigation as prophylaxis against HIV in high-risk women because of its unique pharmacological profile. In addition to the convenience of being a once daily single tablet, TDF's safety profile is comparable to placebo among HIV infected persons, it has striking anti-HIV potency, and it has low potential for selection of resistant viruses. TDF is cleared from the body by the kidneys and is not metabolized by the liver. Therefore, TDF has limited potential to have pharmacokinetic interactions with other hepatically metabolized drugs. Each of these properties is necessary given the realities of the intended target populations. Moreover, initial prevention studies in simian models have provided encouraging results. Finally, the drug's sponsor is supportive of investigating the potential use of TDF as a preventive, as well as a therapeutic agent.

Participants' HIV status is monitored monthly. Participants are also monitored for safety using periodic physical examinations, serial laboratory tests and adverse event queries. Lab tests for kidney and liver function were to be conducted at screening, months 1, 3 and every 3 months thereafter or at the final visit if early withdrawal. To minimize the risk of contracting HIV infection, participants are counseled monthly to use male condoms for each act of intercourse. Participants converting for antibodies to HIV are counseled and referred to medical services as appropriate for each country.

ELIGIBILITY:
Inclusion Criteria:

* HIV seronegative
* Willing and able to give informed consent
* 18 years to 35 years old, inclusive
* Sexually active (on average, coitus 3 times per week)
* Have had more than three sexual partners in the last month
* Willing to use study product as directed
* Willing to adhere to follow-up schedule
* Willing to participate in the study for up to 12 months
* Not pregnant, breast feeding, or desiring a pregnancy during the 12 months of participation
* Have adequate renal function (serum creatinine < 1.5 mg/dL)
* Have adequate liver function (hepatic transaminases [ALT and AST] < 43 U/L)
* Have adequate serum phosphorus (greater than or equal to 2.2 mg/dL)
* In general good health (no active, serious infections that require parenteral antibiotics; no active clinically significant medical conditions, including heart disease, diabetes, asthma, alcoholism, and cancer)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200
Dates: Start 2004-07; Study Completion 2006-03

PRIMARY OUTCOMES:
Effectiveness endpoint is conversion for antibodies to HIV 1 or 2 as determined by an OMT test and confirmed by an ELISA from a finger prick or blood specimen. Discordant results between the OMT and the ELISA will be tested with WB.
Laboratory safety endpoints will include serum creatinine and phosphorus for kidney function, and AST and ALT for hepatic function. Reported adverse events will also be used for clinical evaluation of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Peterson, PhD, Study Director — FHI 360
Locations (3):
- Care and Health Program, Douala, Cameroon
- Virtual Access, Tema, Ghana
- University of College Hospital, Ibadan, Nigeria